CLINICAL TRIAL: NCT07282340
Title: Phentermine's Impact on Treatment in Teens (PhITT): A Randomized Placebo-Controlled Trial of Phentermine for Adolescents With Obesity
Brief Title: Phentermine's Impact on Treatment in Teens
Acronym: PhITT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Russell McCulloh, MD (Network)
Collaborators: National Institutes of Health (NIH) (NIH); IDeA States Pediatric Clinical Trials Network (Network)
Responsible Party: Sponsor-Investigator, Russell McCulloh, MD, Associate Vice chancellor for Clinical Research, UNMC, Heartland DCOC
Organization: Heartland DCOC (Network)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00161879; U24OD038400 (NIH)
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Childhood Obesity
Keywords: Adolescent Obesity; Pediatric Obesity; Weight Loss; BMI Reduction; Phentermine
MeSH Terms: conditions — Pediatric Obesity; Weight Loss | interventions — Phentermine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 2:1 ratio to receive either phentermine 16 mg or placebo once daily for 52 weeks. The study uses a parallel assignment model, where each participant remains in their assigned group throughout the trial. Site-level assignment of treatments to participants will be balanced with respect to sex using a stratified permuted block of varying block size. The study is double-blinded, with participants, investigators, and study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants, care providers, investigators, and outcomes assessors are blinded to treatment assignment. Only the site pharmacist is unblinded to facilitate dispensing of phentermine or placebo. Randomization is centralized and stratified by sex using a permuted block design. Blinding is maintained throughout the study unless unblinding is required for safety reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentermine 16 mg Group (Experimental): Participants in this arm will receive phentermine 16 mg daily, administered as two 8 mg tablets taken orally once
  Interventions: Drug: Phentermine
- Placebo Group (Placebo Comparator): Participants in this arm will receive placebo tablets that are visually identical to the phentermine tablets but contain no active pharmaceutical ingredient. The placebo will be taken orally once daily in the morning for 52 weeks. All participants will also receive lifestyle education handouts at each study visit. This arm serves as the control group for evaluating the efficacy and safety of phentermine in adolescents with obesity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phentermine — Phentermine 16 mg administered orally once daily in the morning for 52 weeks. The dose is provided as two 8 mg tablets. Participants also receive lifestyle education handouts at each study visit. The intervention is designed to evaluate the efficacy and safety of phentermine for weight loss in adolescents with obesity.
  Arms: Phentermine 16 mg Group
Drug: Placebo — Placebo tablets that are visually identical to phentermine tablets but contain no active pharmaceutical ingredient. Administered orally once daily in the morning for 52 weeks. Participants also receive lifestyle education handouts at each study visit. This control arm is used to evaluate the efficacy and safety of phentermine in adolescents with obesity.
  Arms: Placebo Group

SUMMARY:
PhITT is a Phase IIb, multicenter, randomized, double-blind, placebo-controlled clinical trial evaluating the efficacy and safety of phentermine (16 mg daily) in adolescents aged 12 to <18 years with obesity. Conducted across approximately 10 sites within the IDeA States Pediatric Clinical Trials Network (ISPCTN), the study aims to enroll up to 240 participants and then randomize up to 198 who meet eligibility criteria, randomized in a 2:1 ratio to phentermine or placebo over a 52-week treatment period, followed by a 2-week withdrawal assessment.

ELIGIBILITY:
Inclusion criteria* include, but are not limited to:

* Age ≥ 12 years and < 18 years at time of consent;
* Tanner Staging ≥ 2 at the time of screening;
* Obesity (BMI ≥ 95th age- and sex-specific CDC percentile or BMI ≥ 30 kg/m2);
* Biological females must agree to use adequate contraception, defined as double barrier methods, stable hormonal contraception plus single barrier method, tubal ligation, or abstinence.

Exclusion criteria* include, but are not limited to:

* Contraindications to phentermine in adults such as:

  * A history of cardiovascular disease (e.g., coronary artery disease, stroke, clinically significant congenital heart disease, clinically significant cardiac arrhythmias, and congestive heart failure);
  * History of glaucoma;
  * Current or recent (within 14 days of screening) use of a monoamine oxidase (MAO) inhibitor;
  * Any previous history of drug dependency or current use of an illicit substance (positive urine drug screen);
  * Current pregnancy or breastfeeding;
  * Plans to become pregnant within the study duration;
  * Known hypersensitivity to sympathomimetic amines;
* Current nicotine use or nicotine cessation within 3 months of screening;
* Stage 2 hypertension (or greater) or taking any medication to treat hypertension;
* Current type 1 or type 2 diabetes mellitus or taking any medication to treat diabetes or prediabetes;
* Current or recent (within 3 months of screening) use of prescribed weight loss medication(s)/medically prescribed diets (e.g., low calorie, meal replacement/herbal agents/dietary supplements or weight loss program);
* Current or recent (within 3 months of screening) use of other sympathomimetic amines such as stimulants to treat attention- deficit/hyperactive disorder;
* Use of chronic systemic glucocorticoid therapy (consecutive use of 3 months or more) or other steroid hormone therapy other than oral contraceptives;
* Use of tricyclic antidepressants, lithium, levodopa, or dopamine receptor agonists;
* History of bariatric surgery;
* History or current diagnosis of schizophrenia, psychosis, bipolar disorder, or mental illness requiring hospitalization within 12 months of screening;
* History of suicide attempt within 2 years or self-harm within 3 months of screening;
* Current Patient Health Questionnaire-9 (PHQ-9) score of ≥ 10;
* Current suicidal ideation type 4 or 5 on Columbia Suicide Severity Rating Scale (C-SSRS);
* Current Eating Attitudes Test-26 (EAT-26) score ≥ 20 or any history of anorexia or bulimia.
* Current condition or disease interfering with metabolism, such as untreated hypo- or hyperthyroidism, Cushing's syndrome;
* Current clinically significant hepatic aspartate transaminase (AST) or alanine transaminase (ALT) > 3x upper limit of age- and sex-specific normal range or renal disease (creatinine clearance < 60 mL/minute); hypertriglyceridemia (triglyceride ≥ 400 mg/dL) or syndromic or monogenic obesity;
* Any clinically significant abnormalities on a standard 12-lead electrocardiogram at baseline;
* Heart rate > 100 bpm at screening;
* Current or recent use of any investigational medication or device or participation in an interventional clinical trial within 30 days of screening;
* Any clinically significant medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation, investigational product administration, or interpretation of trial results.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in BMI from Baseline at Week 52 | 52 weeks
  Change in body mass index (BMI) expressed as a percentage of baseline BMI at week 52.

SECONDARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (TEAEs) | 52 weeks
  Count of TEAEs deemed probably or definitely related to study drug, including common side effects
Number of Treatment-Emergent Adverse Events of Special Interest (TEAESIs) | 52 weeks
  Count of TEAESIs deemed probably or definitely related to study drug, including tachycardia, hypertension, depression, suicidality, and withdrawal symptoms

OTHER OUTCOMES:
Changes in Cardiometabolic Risk Factor Waist Circumference | 52 weeks
  Change in waist circumference from baseline
Changes in Cardiometabolic Risk Factor Blood Pressure | 52 weeks
  Change blood pressure from baseline
Changes in Cardiometabolic Risk Factor Glucose | 52 weeks
  Change in glucose from baseline
Changes in Cardiometabolic Risk Factor Lipids | 52 weeks
  Change in lipids from baseline
Changes in Cardiometabolic Risk Factor Hemoglobin A1C | 52 weeks
  Change in hemoglobin A1C from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Russell McCulloh, MD, Study Director — UNMC

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data including baseline characteristics, outcome measures and adverse events.
Supporting Information: Study Protocol, SAP, ICF